CLINICAL TRIAL: NCT07287579
Title: Comparison Between Platelet Rich Plasma and Nanofat as an Adjuvant Therapy in Hair Transplantation in Male Androgenic Alopecia
Brief Title: Comparison Between Platelet Rich Plasma and Nanofat as an Adjuvant Therapy in HairTransplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shenoda Gamel Fayez, Assistant lecturer in plastic surgery department, faculty of medicine Sohag University hospital., Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med--25-11-1MD
Record Dates: First submitted 2025-11-22; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Androgenic Alopecia
Keywords: hair transplantation
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group a (Experimental): hair transplantation done alone without platelet rich plasma or nanofat injection
  Interventions: Procedure: hair transplantation
- group b (Experimental): we do injection of platelet rich plasma with hair transplantation
  Interventions: Procedure: hair transplantation
- group c (Experimental): we do injection of nanofat with hair transplantation
  Interventions: Procedure: hair transplantation

INTERVENTIONS:
Procedure: hair transplantation — we compare the effect of nanofat injection and platelet rich plasma in hair transplantation in male androgenic alopecia
  Other Names: hair transplantation with platelet rich plasma; hair transplantation with nanofat injection

SUMMARY:
* To compare the efficacy of platlet rich plasma and Nanofat injection as adjuvant therapies with FUE hair transplantation in improving graft survival rate,
* To measure hair density and thickness postoperatively using dermoscopy or trichoscopy.
* To evaluate patient satisfaction and photographic assessment by blinded evaluators.
* To assess any adverse effects or complications related to each modality

DETAILED DESCRIPTION:
* Ideal candidates for hair transplantation typically present with a clear, stable pattern of hair loss, characterized by at least 50% thinning or balding in 1 or more areas. The scalp must be healthy, with donor hair of good quality and quantity. Patients must have realistic expectations and be free of medical conditions that compromise surgical outcomes. The safe donor zone is located in the mid-occipital region between the upper and lower occipital protuberances, typically containing 65 to 85 follicular units/cm²
* Intra-operative injection of PRP is beneficial in giving faster density, reducing the catagen loss of transplanted hair, early recovery of the skin, the faster appearance of new anagen hair in FUE hair transplantation.
* This study compares the effects of PRP and Nano fat as adjuvants in Androgenic alopecia patients undergoing FUE hair transplantation.
* Nanofat contain stem cells supposed to improve the results of FUE hair transplantation , but the question that we hope to answer at the end of our study which one we recommend as an adjuvant therapy PRP or Nano fat?

ELIGIBILITY:
Inclusion Criteria:

* 1. Male patients with stable androgenic alopecia more than 2 years. 2. Age 20-50 years 3. No recent medical hair loss treatments.

Exclusion Criteria:

* 1. Active scalp infections or scarring alopecia. 2. Systemic diseases affecting wound healing. 3. Platelet disorders or anticoagulant use. 4. Smoking or heavy alcohol intake

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
• To measure hair density using dermoscopy. | • All patients will be followed up about 6-12 months postoperative.
  To measure how many hair follicles in each cubic centimetre

CONTACTS AND LOCATIONS:
Overall Officials: samia saied, MD, Study Chair — Sohag University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evin N, Guray Evin S. Camouflage of Postburn Scarring Alopecia Using Nanofat Grafting and Follicular Unit Hair Transplantation. Plast Reconstr Surg. 2024 Jul 1;154(1):207-215. doi: 10.1097/PRS.0000000000010759. Epub 2023 May 26. PMID 37253046
- See also: Outcome of Intra-operative Injected Platelet-rich Plasma Therapy During Follicular Unit Extraction Hair Transplant: A Prospective Randomised Study in Forty Patients — https://pubmed.ncbi.nlm.nih.gov/27761085/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-11): https://cdn.clinicaltrials.gov/large-docs/79/NCT07287579/Prot_SAP_000.pdf